CLINICAL TRIAL: NCT02384928
Title: Effects of Shinbaro Pharmacopuncture in Sciatic Pain Patients With Lumbar Disc Herniation: a Three-armed, Randomized, Double-blind Controlled Pilot Study
Brief Title: Effects of Shinbaro Pharmacopuncture in Sciatic Pain Patients With Lumbar Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JS-CT-2015-03
Record Dates: First submitted 2015-02-27; First posted 2015-03-10 (Estimated); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Sciatica; Intervertebral Disc Displacement
Keywords: Acupuncture; Pharmacopuncture; Usual Care
MeSH Terms: conditions — Sciatica; Intervertebral Disc Displacement | interventions — Acupuncture Therapy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Shinbaro pharmacopuncture group (Experimental): The Shinbaro pharmacopuncture group will receive 8 interventional sessions of Shinbaro pharmacopuncture at one Hyeopcheok (Huatuo Jiaji, EX B2) point and acupuncture at 5 acupoints (GB30, BL40, BL25, BL23, GB34) 2 times/week over 4 weeks. All groups will take 4 educational program sessions supervised by physicians once a week.
  Interventions: Procedure: Shinbaro pharmacopuncture; Device: Acupuncture; Behavioral: Educational program
- Acupuncture group (Active Comparator): The acupuncture group will receive 8 interventional sessions of acupuncture at one Hyeopcheok (Huatuo Jiaji, EX B2) point and 5 other acupoints (GB30, BL40, BL25, BL23, GB34) 2 times/week over 4 weeks. All groups will take 4 educational program sessions supervised by physicians once a week.
  Interventions: Device: Acupuncture; Behavioral: Educational program
- Usual care group (Active Comparator): The usual care group will receive conventional medicine 2 times/day and 2 sessions/week of physical therapy over 4 weeks. Conventional drugs will be prescribed in an individually-tailored, pragmatic method with reference to most frequently used treatments in patients with a primary diagnosis of LDH (KCD disease classification: M51, M541) according to Korean Health Insurance Review and Assessment (HIRA) 2011 statistics, which include aceclofenac, tramadol hydrochloride, talniflumate, diclofenac sodium, and loxoprofen sodium. All groups will take 4 educational program sessions supervised by physicians once a week.
  Interventions: Drug: Conventional medicine; Procedure: Physical therapy; Behavioral: Educational program

INTERVENTIONS:
Procedure: Shinbaro pharmacopuncture — Pharmacopuncture is a treatment that combines 2 of the most frequented Korean medicine treatment methods - traditional acupuncture and herbal medicine - by injecting herbal medicine extract at acupoints. One Hyeopcheok (Huatuo Jiaji, EX B2) acupoint most relevant to patient symptoms with reference to MRI will be administered Shinbaro pharmacopuncture.
  Arms: Shinbaro pharmacopuncture group
Device: Acupuncture — Five acupoints will be needled to about 1cm depth assisted by an acupuncture guide tube with no manual stimulation such as twirling or lifting and thrusting.
  Arms: Acupuncture group; Shinbaro pharmacopuncture group
Drug: Conventional medicine — Conventional drugs will be prescribed in an individually-tailored, pragmatic method with reference to most frequently used treatments in patients with a primary diagnosis of LDH (KCD disease classification: M51, M541) according to Korean Health Insurance Review and Assessment (HIRA) 2011 statistics. The most frequently prescribed conventional drugs for LDH include aceclofenac (Drug class: nonsteroidal antiinflammatoy drugs (NSAIDs)), tramadol hydrochloride (Drug class: Opioids), talniflumate (Drug class: NSAIDs), diclofenac sodium (Drug class: NSAIDs), and loxoprofen sodium (Drug class: NSAIDs).
  Other Names: Conventional drugs
  Arms: Usual care group
Procedure: Physical therapy — Physical therapy will be prescribed with reference to most frequently used treatments in patients with a primary diagnosis of LDH (KCD disease classification: M51, M541) according to Korean Health Insurance Review and Assessment (HIRA) 2011 statistics.
  Other Names: Physiotherapy
  Arms: Usual care group
Behavioral: Educational program — Educational program sessions supervised by physicians will be provided once a week for 4 weeks.The education program will inform the patient of the favorable prognosis of LDH, and instructions for everyday activities and self-management. The education program will consist of handbooks handed out to each participant, and weekly reminders and encouragement from the physician.

SUMMARY:
This trial will evaluate the comparative clinical effectiveness of pharmacopuncture for severe non-acute sciatic pain patients diagnosed with lumbar disc herniation (LDH) with usual care of conventional medicine and that of Korean medicine (acupuncture). Sixty patients with severe non-acute sciatic pain patients diagnosed with LDH (NRS ≥5, 4 weeks - 6 months) will be recruited, and randomized 20 each to the Shinbaro pharmacopuncture, acupuncture, and usual care group, respectively. The 2 acupuncture groups will receive 2 sessions/week of acupuncture alone or with pharmacopuncture for 4 weeks, and the usual care group will receive conventional medication 2 times/day and 2 sessions/week of physical therapy. Post-treatment evaluations will take place 5, 7, 9, and 12 weeks after randomization.

DETAILED DESCRIPTION:
This study is a three-armed, randomized, patient, physician, and assessor-blinded, controlled pilot to the aim of evaluating the comparative clinical effectiveness of pharmacopuncture for severe non-acute sciatic pain patients diagnosed with lumbar disc herniation (LDH) with usual care of conventional medicine and that of Korean medicine (acupuncture). Sixty patients with severe non-acute sciatic pain patients diagnosed with LDH (NRS ≥5, onset between 4 weeks and 6 months) will be recruited, and randomized 20 each to the Shinbaro pharmacopuncture (pharmacopuncture+acupuncture), acupuncture, and usual care group, respectively. The 2 acupuncture groups will receive 2 sessions/week of acupuncture alone or with pharmacopuncture for 4 weeks (total 8 sessions), and the usual care group will receive conventional medication 2 times/day and 2 sessions/week of physical therapy (total 8 sessions). The initial acupuncture physician will administer acupuncture at 5 acupoints (GB30, BL40, BL25, BL23, GB34) in the 2 acupuncture groups, and mark an additional acupoint. A second acupuncture physician will administer pharmacopuncture to the marked acupoint in the pharmacopuncture group, and acupuncture in the acupuncture group. Post-treatment evaluations will take place 5, 7, 9, and 12 weeks after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Sciatica patients with an average sciatic pain NRS of 5 or higher during the preceding 3 days
* Onset of at least 4 weeks previous for current sciatic pain episode
* Patients whose sciatic symptoms correlate with the LDH confirmed on MRI
* Patients who have agreed to follow the trial protocol

Exclusion Criteria:

* Patients who have received invasive treatments such as nerve blocks, pharmacopuncture, or acupuncture within the past week
* Non-spinal or soft tissue pathologies which may cause LBP or sciatic pain (e.g. spinal tumors, rheumatic arthritis)
* Pregnancy
* History of spinal surgery, or spinal pathologies other than LDH (e.g. spinal dislocation, fracture)
* Severe progressive neurologic symptoms (e.g. cauda equina syndrome, progressive muscle weakness)
* Patients for whom acupuncture may be inappropriate or unsafe (e.g. hemorrhagic diseases, blood clotting disorders, history of anti-coagulation medicine, severe diabetes with risk of infection, severe cardiovascular diseases or other conditions deemed unsuitable)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09-09 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-03-16 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) of sciatic pain | Week 5
  On the 10cm line which represent the severity of pain, the patient mark point which best represent the severity that he feels.

SECONDARY OUTCOMES:
Visual analogue scale (VAS) of sciatic pain | Week 1, 2, 3, 4, 7, 9, 12
  On the 10cm line which represent the severity of pain, the patient mark point which best represent the severity that he feels.
Visual analogue scale (VAS) of low back pain (LBP) | Week 1, 2, 3, 4, 5, 7, 9, 12
  On the 10cm line which represent the severity of pain, the patient mark point which best represent the severity that he feels.
Numeric rating scale (NRS) of low back pain (LBP) | Baseline(screening), Week 1, 2, 3, 4, 5, 7, 9, 12
  The patient choose number between 0 to 10, which represent the serverity of the pain that he felt. 0 means there's no pain, and 10 means there's severe pain that he ever felt.
Numeric rating scale (NRS) of sciatic pain | Baseline(screening), Week 1, 2, 3, 4, 5, 7, 9, 12
  The patient choose number between 0 to 10, which represent the serverity of the pain that he felt. 0 means there's no pain, and 10 means there's severe pain that he ever felt.
Oswestry Disability Index (ODI) | Week 1, 2, 3, 4, 5, 7, 9, 12
  The Oswestry Disability Index (ODI) is an index is derived from the Oswestry Low Back Pain Questionnaire used by clinicians and researchers to quantify disability for low back pain. The ODI is a 10-item score from 0 to 100 that encompasses limitations in activity, sleeping, social life, work, and personal care resulting from low back pain.
Short Form Health Survey 36 (SF-36) | Week 1, 5, 7, 12
  SF-36 Questionnaire consists of several questions related to local pain, radiationg pain, analgesic intake and ability.
EuroQol-5 Dimension (EQ-5D) | Week 1, 5, 7, 12
  Estimates that shows the quality of life(QOL).
Patient Global Impression of Change (PGIC) | Week 1, 5, 7, 12
  This scale evaluates all aspects of patients' health and assesses if there has been an improvement or decline in clinical status.
Number and percentage of participants with adverse events | Week 1, 2, 3, 4, 5, 7, 9, 12
  The number and percentage of participants with adverse events, categorized by affected body region, will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Jinho Lee, Principal Investigator — Jaseng Medical Foundation
Locations (1):
- Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee J, Shin JS, Lee YJ, Kim MR, Ahn YJ, Park KB, Kropf MA, Shin BC, Lee MS, Ha IH. Effects of Shinbaro pharmacopuncture in sciatic pain patients with lumbar disc herniation: study protocol for a randomized controlled trial. Trials. 2015 Oct 12;16:455. doi: 10.1186/s13063-015-0993-6. PMID 26459006